CLINICAL TRIAL: NCT03479593
Title: Identification of Culprit Lesions in Non ST-elevation Myocardial Infarction and Multivessel Disease
Brief Title: Culprit Lesions in NSTEMI With Multi Vessel Disease (NSTEMI-CULPRIT)
Acronym: NS-CULPRIT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Thomas Engstrom, Professor, Rigshospitalet, Denmark
Other Study IDs: H-17023377
Record Dates: First submitted 2017-11-27; First posted 2018-03-27 (Actual); Last update posted 2023-03-29 (Actual); Status verified 2023-03

CONDITIONS: NSTEMI - Non-ST Segment Elevation MI; Multi Vessel Coronary Artery Disease
Keywords: NSTEMI; Culprit; Cardiac magnetic resonance; Optical Coherence Tomography
MeSH Terms: conditions — Non-ST Elevated Myocardial Infarction | interventions — Tomography, Optical Coherence; Microvascular Density

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- CMR and OCT in NSTEMI patients with MVD: NSTEMI patients with multi vessel disease
  Interventions: Diagnostic Test: CMR and OCT in NSTEMI patients with MVD

INTERVENTIONS:
Diagnostic Test: CMR and OCT in NSTEMI patients with MVD — Lesions >50% stenosis i patients with NSTEMI are examined by OCT. All patients will have CMR performed prior to angiography

SUMMARY:
Acute myocardial infarction owes to a plaque rupture resulting in total (STEMI) or partial occlusion (NSTEMI) of the coronary artery. In patients with a partial occlusion and multi vessel disease (MVD), identification of the lesion responsible for the current event (culprit) at the time of the examination (coronary angiogram, CAG) can be difficult.

Meanwhile, identification of the culprit lesion is vital to conduct proper treatment. Furthermore, treating an artery with no plaque rupture (non-culprit), imposes a small risk for complications, which may be fatal. Precise identification of the culprit lesion in NSTEMI patients with MVD remains unsettled

The purpose of this study is proper and precise identification of the culprit lesion in NSTEMI patients with MVD.

DETAILED DESCRIPTION:
Background

Acute myocardial infarction owes to a plaque rupture resulting in total (STEMI) or partial occlusion (NSTEMI) of the coronary artery. Current guidelines in NSTEMI recommend an invasive coronary angiogram (CAG) and possible treatment with percutaneous intervention (PCI) within 2-72 hours. In NSTEMI patients and multi vessel disease (MVD), identification of the lesion responsible for the current event (culprit) at the time of the examination can be difficult.

Meanwhile, identification of the culprit lesion is vital to conduct proper treatment in order to restore blood flow to the myocardium. Furthermore, treating an artery with no plaque rupture (non-culprit), imposes a small risk for complications, which may be fatal. In addition, since the symptoms relate to the culprit lesion it is currently unclear whether all stenosis or only the culprit should be treated by PCI. Today precise identification of the culprit lesion in NSTEMI patients with MVD remains unsettled.

Purpose

The overall objective of this study is proper and precise identification of the culprit lesion in NSTEMI patients with MVD.

Methods

The study employs cardiac magnetic resonance (CMR), which allows detection of myocardium exposed to even brief periods of ischemia. Furthermore, Optical Coherence Tomography (OCT) which visualises the coronary artery lumen and wall. OCT allows for direct visualization of atherosclerotic plaques, presence of thrombus and atherosclerotic plaque ruptured that cannot be seen on a CAG alone.

Patients will have CMR performed prior to CAG. The PCI operator determines culprit based on CAG and ECG changes alone. OCT is subsequently performed on culprit lesion(s) and stenosis ≥ 50%.

Sample size calculation

Assuming the culprit lesion can be correctly identified with history/angiography/ECG in 95% of cases a positive predictive value >90% with 95% accuracy can be reached with 100 patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients > 18 years of age
* NSTEMI (ECG changes and/or troponin/creatine kinase myocardial band (CK-MB) rise) within 48 hours after symptom debut.
* Multivessel disease at CAG: More than one vessel with >50% stenosis.

Exclusion Criteria:

* Known intolerance of heparin or contrast medium.
* Inability to understand information or to provide informed consent.
* estimated glomerular filtration rate (eGFR) < 30 ml/min.
* Other reasons for troponin rise not applicable to acute myocardial infarction.
* Atrial fibrillation at admission.
* Patients with contraindication for CMR will only have OCT performed.
* Potential pregnancy
* Unstable patients requiring acute CAG and PCI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligible NSTEMI patients scheduled for CAG at one center
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2018-01-10 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2024-01-01 (Estimated)

PRIMARY OUTCOMES:
Is the PCI operator capable of identifying the culprit lesion based on ECG-changes and CAG? (CMR is the golden standard) | Through study completion, an average of 1 year
  Correlation between operator identification of the culprit and CMR/OCT. The location of the culprit on CAG/ECG and OCT versus CMR will be evaluated by the chi2-test

SECONDARY OUTCOMES:
Positive predictive value of PCI operator identification of culprit lesion with CAG and ECG. | Through study completion, an average of 1 year
  cross-tables will be used to calculate the positive predictive value Receiver-operating-characteristics will be used to compare the additional diagnostic value of OCT compared to CAG/ECG.
Improvement in identification of culprit lesions evaluated by identification of an additional diagnostic value of OCT compared to CAG/ECG | Through study completion, an average of 1 year
  Receiver-operating-characteristics will be used to compare the additional diagnostic value of OCT compared to CAG/ECG. CMR is the golden standard.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Engstrøm, DMSCi, PhD, Principal Investigator — Rigshospitalet, University of Copenhagen
Locations (1):
- Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No